CLINICAL TRIAL: NCT04184089
Title: High Flow Nasal Cannula in Patients Undergoing Endoscopic Retrograde Cholangiopancreatography With Intravenous Sedation.
Brief Title: High Flow Nasal Cannula in Patients Undergoing ERCP Retrograde Cholangiopancreatography With Intravenous Sedation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Christian Rouphael, Instructor of Clinical Specialty, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANES.CE.01
Record Dates: First submitted 2019-10-11; First posted 2019-12-03 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: High-flow Nasal Cannula; Intravenous Sedation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Experimental): High flow rate of 5 L/min and FiO2 of 40%
  Interventions: Device: High flow nasal cannula (15 L/m)
- Group 15 liter (Experimental): Nasal cannula at flow rate of 15 L/min and FiO2 of 40%
  Interventions: Device: High flow nasal cannula (30 L/m)
- Group 60 liter (Experimental): Nasal cannula at flow rate of 60 L/min and FiO2 of 40%
  Interventions: Device: High flow nasal cannula (60 L/m)

INTERVENTIONS:
Device: High flow nasal cannula (15 L/m) — nasal cannula at a flow rate of 15 l/min and FiO2 of 40%
  Arms: Control group
Device: High flow nasal cannula (30 L/m) — nasal cannula at a flow rate of 30l/min and FiO2 of 40%
  Arms: Group 15 liter
Device: High flow nasal cannula (60 L/m) — nasal cannula at flow rate of 60L/min. Oxygen supplementation will be at an FiO2 of 40%.
  Arms: Group 60 liter

SUMMARY:
The aim of the current study is to compare the incidence of oxygen desaturation in patients receiving HFNC at different flow rates compared to conventional oxygen therapy via a simple cannula during ERCP. Secondary outcomes include lowest average observed oxygen saturation (SpO2), snoring classification scores and satisfaction levels of both patients and gastroenterologists.

Participants will be randomized to 3 groups: G0 will receive a 5 l/ min flow rate through a nasal cannula at and FiO2 of 40 %, G1 will receive a 15 l/ min flow rate and FiO2 of 40% and G2: will receive a 60L/min flow rate and FiO2 of 40%.

DETAILED DESCRIPTION:
High flow nasal cannula provides adequate oxygenation in patients with compromised pulmonary function. Very few studies in the literature addressed its use with IV sedation in the OR. Successful application of High Flow nasal cannula in intravenous deep sedation cases in the OR will benefit in the reduction of airway manipulation and side effects from general anesthesia.

The aim of the current study is to compare the incidence of oxygen desaturation in patients receiving HFNC at different flow rates compared to conventional oxygen therapy via a simple cannula during ERCP. Secondary outcomes include lowest average observed oxygen saturation (SpO2), snoring classification scores and satisfaction levels of both patients and gastroenterologists.

A total of 60 patients undergoing ERCP will be equally randomized to 3 groups:

G0: will receive a 5 l/ min flow rate through a nasal cannula at and FiO2 of 40 %, G1: will receive a 15 l/ min flow rate and FiO2 of 40% and G2: will receive a 60L/min flow rate and FiO2 of 40%.

The three groups' intra-procedure and outcome parameters and variables will be compared. Statistical comparison will be made using the ANOVA, Student's t-test, and Chi-squared test. Level of statistical significance will be considered at p<0.05. ANOVA test will be performed to compare the different means between the four groups. Minimum and maximum 3 of 17 values will be recorded for each value in all 3 groups. A two sided P value of less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Patient able to give consent.
2. Patient undergoing deep sedation.
3. Patient undergoing ERCP procedure with no restrictions on the duration of the procedure.
4. Age > 18 years
5. Patients with BMI < 40 kg/m2

Exclusion Criteria:

1. Patient unable to give consent
2. Patient refusal to participate
3. Patients undergoing general anesthesia
4. age less than 18 years old
5. Patients with severe heart failure (EF<30%)
6. Morbidly obese Patients with BMI > 40 kg/m2
7. Patients with sleep apnea
8. Claustrophobia
9. Risk of aspiration due to severe reflux
10. Facial injury, facial malformation
11. Nasal defects/obstruction
12. ASA 4 patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
Desaturation | During the surgery
  Desaturation (SpO2≤95%) or a drop of more than 5% from baseline SpO2

SECONDARY OUTCOMES:
Lowest SpO2 | During procedure
  Lowest SpO2 (%)
Mean SpO2 | During procedure
  Mean SpO2 (%)
Duration of the procedure | During procedure
  Duration of the procedure measured in minutes
Snoring status | During procedure
  Snoring status measured as Yes/No
Snoring snore | During procedure
  snoring score assessed using a subjective snoring classification developed at Stanford on a scale from 0 to 10
Gastroenterologists' satisfaction | During procedure
  Gastroenterologists' satisfaction measured using a 5-point Likert scale
Patients' satisfaction | During procedure
  Patients' satisfaction measured using a 5-point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Christian Rouphael, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- Christian Rouphael, Beirut, Lebanon